CLINICAL TRIAL: NCT04142294
Title: Safety of Graded-Dose of Histidine as Determined by Circulating Analytes, Sleep Records, Physical Activity, Anthropometric Measurements, and Mood
Brief Title: Safety of Graded-Dose of Histidine in Humans
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cornell University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Other
Other Study IDs: 83676/A001
Record Dates: First submitted 2018-10-30; First posted 2019-10-29 (Actual); Last update posted 2022-02-07 (Actual); Status verified 2022-01

CONDITIONS: Healthy
MeSH Terms: interventions — Histidine

STUDY DESIGN:
Intervention Model Description: Histidine supplementation trial, non-randomized, sequential delivery of graded doses of the amino acid histidine. All participants serve as their own controls. Following baseline measurements, subjects ingest encapsulated high quality histidine for four continuous weeks at graded doses of 4, 8 and 12 g/day. A forth dose at 16 g/day is assessed if no adverse outcomes are observed for the three graded doses. Histidine doses are suggested based on experience with other amino acids (relative difference of average intake and metabolic limits). Each dose is followed by a 3-week minimum recovery period. During the recovery period, subjects will continue to be monitored (vitals and weight) but no supplementation is consumed. At the conclusion of each washout period, before the start of the next dose, subjects provide a blood sample, vitals (blood pressure and heart rate), weight, 4-day diet record, sleep log, hunger and satiety VAS, mood VAS, and physical activity monitoring.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- 4 g / day histidine (Experimental): subjects ingest encapsulated high quality histidine for four continuous weeks at 4 g/day.
  Interventions: Dietary Supplement: Histidine
- 8 g / day histidine (Experimental): subjects ingest encapsulated high quality histidine for four continuous weeks at 8 g/day
  Interventions: Dietary Supplement: Histidine
- 12 g /day histidine (Experimental): subjects ingest encapsulated high quality histidine for four continuous weeks at 12 g/day
  Interventions: Dietary Supplement: Histidine
- 16 g /day histidine (Experimental): subjects ingest encapsulated high quality histidine for four continuous weeks at 16 g/day. The 16 g /day dose will be administered if no adverse effects are observed for doses 4-12 g/day
  Interventions: Dietary Supplement: Histidine

INTERVENTIONS:
Dietary Supplement: Histidine — ingestion of encapsulated high quality histidine for four continuous weeks followed by a washout period of 3 weeks

SUMMARY:
Histidine is an essential amino acid with health benefits that include anti-inflammatory, anti-oxidant, glucoregulatory, and weight management. The current expert opinion for histidine intake is 8 and 12 mg/(kg body weight per day), an estimate that was extrapolated from the infant requirement for histidine. Further, the clinical safety of histidine supplementation above the average dietary intake has not been determined.The overarching objectives are to 1) measure the safety of histidine supplementation and 2) measure the potential benefits of histidine at doses above the average intake and current recommendation in a healthy adult population.

DETAILED DESCRIPTION:
Histidine is an essential amino acid with health benefits that include anti-inflammatory, anti-oxidant, glucoregulatory, and weight management. Because of the extended period of time (>35 days) that is required to deplete body histidine pools in adults, it has not been possible to fully determine histidine requirements. The current expert opinion for histidine intake is 8 and 12 mg/(kg body weight per day), an estimate that was extrapolated from the infant requirement for histidine. The average intake of histidine from a normal adult diet in the U.S., Europe, and Japan was reported between 2.12 and 2.40 g/day with the 99th percentile intake in men at 50-70 years of age consuming 5.20 g/day. The clinical safety of histidine supplementation above the average dietary intake has not been determined. Therefore, this study will utilize graded doses of histidine that are at are moderately above the average intake to identify safety and benefits of histidine in a healthy human population. Further, the clinical safety of histidine supplementation above the average dietary intake has not been determined.The overarching objectives are to 1) measure the safety of histidine supplementation and 2) measure the potential benefits of histidine at doses above the average intake and current recommendation in a healthy adult population. Following the completion and review of a health history questionnaire, vitals, and a biochemical panel, participants will be deemed healthy by a nurse practitioner and able to participate. After baseline measures are obtained, supplements (encapsulated histidine) will be provided at three graded doses (4 g/day, 8 g/day and 12 g/day) a forth dose (16 g/day) will be consumed if no adverse effects are observed at the three graded doses. Each dose will be for 28 days followed by a three week recovery period. At baseline, weeks 2 and 4 of supplement, and recovery a basic biochemical panel, anthropometric, urinary and serum zinc, will be conducted. Additionally, body composition will be conducted at baseline and week 4 of each dose. Changes in dietary intake and physical activity will be measured with 4-day food records and Actigraph activity monitors, respectively. Changes in sleep patterns will be measured with the Pittsburgh sleep questionnaire.

ELIGIBILITY:
Inclusion Criteria:

• healthy young males and females aged 21-50 y.

Exclusion Criteria:

* A body-mass index (BMI) <19.9 kg/m2 or > 29.9 kg/m2
* taking/on immunosuppressive medications or prescription anti-coagulation therapy
* pregnancy
* breastfeeding
* musculoskeletal disorder
* diabetes
* alcoholism (>11 drinks per week for women, >14 drinks per week for men) or other drug addiction
* acute illness
* inability to travel to Cornell University campus
* A blood pressure at or above 140/90
* For individuals desiring to participate in the optional biopsy, a history of a negative or allergic reaction to local anesthetic is an exclusion criteria

Ages: 21 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2017-09-21 (Actual); Primary Completion 2019-08-31 (Actual); Study Completion 2019-08-31 (Actual)

PRIMARY OUTCOMES:
Change in concentration of zinc in mg/ml | at week 0 and 4 of each dose
  The safety of histidine supplementation at each dose is monitored through blood markers of zinc
Change in concentration of liver enzymes (ALT, ALP, and AST) in Units per Liter | at weeks 0 (washout), 2 and 4 of each dose
  The safety of histidine supplementation at each dose is monitored through circulating liver enzymes
Change in body weight in kilograms | at weeks 0 (washout), 2 and 4 of each dose
  The safety of histidine supplementation at each dose is monitored through changes in weight
Change in concentration of total protein and albumin in g/dl | at weeks 2 and 4 of each dose
  The safety of histidine supplementation at each dose is monitored through circulating total protein and albumin
Change in concentration of blood urea nitrogen, Creatinine, bilirubin and glucose each in mg/gL | at weeks 0 (washout), 2 and 4 of each dose
  The safety of histidine supplementation at each dose is monitored through circulating blood urea nitrogen, Creatinine, bilirubin and glucose
Change in concentration of C-reactive protein mg/L | at weeks 0 (washout), 2 and 4 of each dose
  The safety of histidine supplementation at each dose is monitored through circulating CRP
HgbA1c in % | at week 4 of each dose
  The safety of histidine supplementation at each dose is monitored through circulating HgbA1c
Change in heart rate in beats per minute | weeks 0 (baseline and washout), 1, 2, 3, and 4 of each dose
  The safety of histidine supplementation at each dose is monitored through heart rate
Change in systolic and diastolic blood pressures in mmHG | weeks 0 (baseline and washout), 1, 2, 3, and 4 of each dose
  The safety of histidine supplementation at each dose is monitored through blood pressure

SECONDARY OUTCOMES:
Change in hours of sleep | week 0 to 4 of each dose
  The effects of histidine will be assessed with changes in sleep pattern as determined using a subjective measurement tool
Change in dietary intake of energy, macronutrients, and amino acids measured in kcals and g/day with 4 day food record | week 0 to 4 of each dose
  The effects of histidine will be assessed with changes dietary intake as determined with 4 day food records
Change in physical activity measured in steps per day | week 0 to 4 of each dose
  The effects of histidine will be assessed with changes in physical activity patterns using an Actigraph
Change in subjective mood measured in arbitrary units | week 0 to 4 of each dose
  The effects of histidine will be assessed with changes in mood as determined using a subjective visual analog scale. 100 mm line is anchored by two opposing statements. The higher number the greater the mood.
Change in subjective desire to eat measured in arbitrary units | week 0 to 4 of each dose
  The effects of histidine will be assessed with changes in desire to eat will be determined using a visual analog scale. 100 mm line is anchored by two opposing statements. The greater the number the stronger the desire.

CONTACTS AND LOCATIONS:
Locations (1):
- Human Metabolic Research Unit, Ithaca, New York, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Gheller ME, Vermeylen F, Handzlik MK, Gheller BJ, Bender E, Metallo C, Aydemir TB, Smriga M, Thalacker-Mercer AE. Tolerance to graded dosages of histidine supplementation in healthy human adults. Am J Clin Nutr. 2020 Nov 11;112(5):1358-1367. doi: 10.1093/ajcn/nqaa210. PMID 32766885